CLINICAL TRIAL: NCT00307385
Title: Modulation of Motor Learning After Stroke Using Principles of Metaplasticity
Brief Title: Transcranial Direct Current Stimulation to Improve Hand Movement in Stroke Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060127; 06-N-0127
Record Dates: First submitted 2006-03-25; First posted 2006-03-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-03-27

CONDITIONS: Stroke
Keywords: Motor Recovery; Transcranial Direct Current Stimulation (tDCS); Homeostatic Plasticity; Ipsilesional Primary Motor Cortex; Paretic Fingers Motor Sequence; Motor Cortex; Motor Function; Motor Learning; Premotor Cortex; Primary Motor Cortex; Stroke; Healthy Volunteer; HV
MeSH Terms: conditions — Stroke

SUMMARY:
This study will examine whether hand movement in stroke patients can be improved by applying electrical stimulation to the side of the brain affected by the stroke. It will compare the effects of similar brain stimulations in stroke patients and healthy volunteers.

Healthy, right-handed normal volunteers and stroke patients between 18 and 80 years of age may be eligible for this study. Patients' stroke must have occurred at least 3 months before entering the study and affect one side of the brain only. Candidates are screened with a medical history, brain MRI, and evaluation of memory and attention span. Pregnant women are excluded from the study.

The study involves seven 2-day sessions over the course of about 8 weeks, with each session separated by at least 1 week. During each session participants practice a pattern of hand movements and their accuracy in performing the movements is evaluated before and after brain electrical stimulation. The movements include a complex finger sequence, a simple finger sequence, a peg test (placing wooden pegs in holes on a board), a hand function test (turning over cards, picking up small objects with one hand and placing them in a can, picking up small objects with a spoon and placing them in a can, stacking checkers, moving light cans, and moving heavy cans), and a box and block test (picking up and moving blocks from one box to another).

The first day of each 2-day session lasts about 5 hours and includes the following:

* TMS measurements: A wire coil is held on the scalp, and a brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. During the stimulation, the subject may be asked to tense certain muscles slightly or perform other simple actions. The stimulation may cause a twitch in muscles of the face, arm, or leg, and the subject may hear a click and feel a pulling sensation on the skin under the coil.
* tDCS: Small, wet sponge electrodes are applied to the head - one above the eye and the other on the back of the head. A small electrical current is passed between them. The subject may feel an itching or tingling sensation under the electrodes or see light flashes. Some sessions are done with sham tDCS.
* Motor learning under tDCS: tDCS is repeated while the subject performs different finger movements. A new pattern of finger movements is taught each session.
* Surface electromyography: Electrodes are filed with a conductive gel and taped to the skin over one small hand muscle to measure the electrical activity of muscles.
* Behavioral measurements: Evaluation of learned movement tasks
* Questionnaires to evaluate the subject's attention, fatigue and mood before and after testing

The second day of each session lasts about 2 hours and includes the TMS measurements and behavior measurements.

DETAILED DESCRIPTION:
Objectives: Recent advances in neuroscience may be helpful in designing more accurate neurorehabilitative strategies to decrease post-stroke disability. First, recovery is more extensive when the interhemispheric balance of activity favors the ipsilesional primary motor (M1Ipsilesional) and premotor (PMIpsilesional) cortices. Second, non-invasive transcranial direct current stimulation (tDCS) over M1Ipsilesional may help to transiently improve motor performance in stroke patients. Third, in healthy volunteers, training combined with cortical stimulation of M1 (which plays a critical role in motor learning) leads to up-regulation of corticomotor excitability, improved motor learning, and use-dependent plasticity. Since stroke patients have to re-learn how to control their paretic hand, enhancing their learning capacity by adequate tuning of M1Ipsilesional with tDCS could promote plastic reorganization that supports functional improvement. Finally, another factor to be considered is that functional changes elicited by cortical stimulation depend on the previous activity state (metaplasticity). Therefore, we hypothesize that implementing metaplastic changes will enhance motor learning gains induced by tDCS in chronic stroke patients to a larger extent than a control intervention in both stroke patients and healthy volunteers.

Study Population: 20 healthy subjects for safety issues and parameter optimization; 31 patients with a single cortical or sub-cortical stroke; and 31 matched healthy controls.

Design: To test our hypothesis, we will precondition M1Ipsilesional with cathodal tDCS (which transiently down-regulates activity in this site) and then apply anodal tDCS to M1Ipsilesional during a motor sequence learning with the paretic hand. After a familiarization session, real and sham tDCS will be applied in 6 randomized sessions in a crossover design. Learning will be evaluated one day after each tDCS/sham session.

The primary outcome measure will be the number of learned sequences correctly played on a keyboard in a 30-second period. TMS will be used 1) to interfere with the activity of different cortical motor areas as a marker of their respective contribution to paretic hand control before and after the metaplasticity intervention and 2) to measure corticomotor excitability changes associated with the interventions. This will provide descriptive information on the neural substrates underlying behavioral gains, important for hypothesis-generation and power analysis in future investigations.

ELIGIBILITY:
* INCLUSION CRITERIA:

Stroke Patients:

* age between 18-80 years
* first-ever, single stroke with thromboembolic non-hemorrhagic hemispheric lesions
* stroke more than 3 months ago
* stroke that affected one side of the brain (unilateral stroke)
* Patients with initially a severe motor paresis (below MRC grade 2), who subsequently recovered to the point that they have a residual motor deficit but can perform the required tasks (i.e., perform relatively independent finger movements)
* willing and able to give consent

Healthy Volunteers:

* age between 18-80 years
* able to perform tasks required by the study
* willing and able to give consent

EXCLUSION CRITERIA:

Stroke Patients:

* unable to perform the tasks of the study
* more than one stroke
* both sides of the brain affected or clear bilateral motor impairment
* stroke in the cerebellum or brainstem
* increased intracranial pressure as evaluated by clinical means
* history of severe alcohol or drug abuse, psychiatric illness like severe depression, poor motivational capacity, or severe language disturbances, particularly of receptive nature or with serious cognitive deficits (defined as equivalent to a mini-mental state exam score (MMSE) of 23 or less), or degenerative brain processes such as Alzheimer's disease
* severe uncontrolled medical problems (e.g., cardiovascular disease, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, or a deteriorated condition due to age, uncontrolled epilepsy or others), more than moderate to severe microangiopathy, polyneuropathy, diabetes mellitus, or ischemic peripheral disease
* receiving drugs acting primarily on the central nervous system, which lower the seizure threshold such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants (for the TMS component)
* pregnant
* medical or technical contraindications to MRI procedures or devices producing artifacts that impair MRI signal (e.g., dental braces, pacemakers, implanted medication pumps, cochlear devices, neural stimulators, metal in the cranium, surgical clips, and other metal/magnetic implants, claustrophobia)

Healthy volunteers:

* unable to perform the tasks
* history of severe alcohol or drug abuse, psychiatric illness like severe depression, poor motivational capacity, or severe language disturbances, particularly of receptive nature or with serious cognitive deficits (defined as equivalent to a mini-mental state exam score (MMSE) of 23 or less), or degenerative brain processes such as Alzheimer's disease
* severe uncontrolled medical problems (e.g., cardiovascular disease, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, or a deteriorated condition due to age, uncontrolled epilepsy or others), more than moderate to severe microangiopathy, polyneuropathy, diabetes mellitus, or ischemic peripheral disease
* problems with movement of the hands
* receiving drugs acting primarily on the central nervous system, which lower the seizure threshold such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants (for the TMS component)
* pregnant
* medical or technical contraindications to MRI procedures or devices producing artifacts that impair MRI signal (e.g., dental braces, pacemakers, implanted medication pumps, cochlear devices, neural stimulators, metal in the cranium, surgical clips, and other metal/magnetic implants, claustrophobia)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82
Dates: Start 2006-03-23; Study Completion 2008-03-27

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Fridman EA, Hanakawa T, Chung M, Hummel F, Leiguarda RC, Cohen LG. Reorganization of the human ipsilesional premotor cortex after stroke. Brain. 2004 Apr;127(Pt 4):747-58. doi: 10.1093/brain/awh082. Epub 2004 Jan 28. PMID 14749291